CLINICAL TRIAL: NCT00246844
Title: Assessing Arginine-Stimulated Native Pancreas Insulin Production Via Selective Venous Sampling in Patients With Long-Functioning Pancreas Allografts
Brief Title: Assessment of Insulin Production From Native Pancreas in Patients With Pancreas Transplants
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060019; 06-DK-0019
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Long-Functioning Pancreas Allografts; Pancreas Transplant
Keywords: Transplant; Diabetes; C-Peptide; B Cell; Immunosuppression; Type 1 Diabetes; Pancreas Transplant
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

SUMMARY:
This study will examine whether insulin-producing cells in the pancreas (beta cells) can recover in patients with type 1 diabetes who have had a pancreas transplant. In type 1 diabetes, the body's immune system destroys the beta cells. Patients are treated with insulin shots or a pancreas transplant to control their blood sugar. Some experiments suggest that the pancreas may have the capacity to recover some of its insulin-producing capacity, but that ability is negated by factors such as the continuing immune attack and erratic blood sugar levels in patients.

Patients who have had a pancreas transplant may be in a unique situation to allow their own pancreas to regrow beta cells for two reasons: 1) the medicines they take to prevent rejection of the transplanted pancreas weaken their immune system; and 2) they have near-normal blood sugar levels because of their functioning transplanted pancreas. This study will test this hypothesis by sampling blood from patients' hepatic vein, which drains the liver and native pancreas and from their iliac vein, which drains the transplanted pancreas. This will determine whether insulin is coming from the transplanted pancreas (iliac vein) or the liver and native pancreas (hepatic vein).

Patients 18 years of age and older who have had stable pancreatic transplant function for more than 5 years may be eligible for this study. Candidates are screened with a medical history and physical examination.

Participants are admitted to the hospital for 2 days for a full medical examination, blood tests and procedures to determine insulin production. The procedures will include the placement of catheters in the neck and groin for blood sampling. Participants will be closely monitored after the procedures and discharged home if there are no complications.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is thought to result from an autoimmune destruction of insulin producing beta-cells found within the pancreatic islets of Langerhans. In addition to the autoimmune process however, many studies have shown that hyperglycemia is also toxic to islets. Interventional studies have shown, for instance, that either tight glycemia control or immunosuppression can preserve C-peptide production. We hypothesize that patients who are immunosuppressed and euglycemic will display evidence that their native pancreas has recovered beta-cell function. We have asked whether pancreas transplant recipients, due to the immunosuppression required to prevent allograft loss, and the improved glycemia control resulting from the transplanted pancreas, might display some recovery of their native pancreatic islet function. Our preliminary data suggest that patients without C-peptide production prior to receiving an islet transplant appear to recover some endogenous pancreatic insulin secretion after islet transplantation. We will study whole pancreas transplant recipients, specifically those with grafts functioning for at least 5 years. We will test for native pancreas insulin production by infusing arginine into a peripheral vein, then selectively/simultaneously sampling blood for C-peptide levels from the hepatic veins and the vein draining the pancreatic allograft . Unlike our previous study of islet transplant recipients, a study that required portal vein cannulation, this study will require only hepatic and iliac vein cannulations, both much easier to accomplish, and associated with much less risk to the patient. Samples obtained from these sites will be tested for C-peptide levels. In addition, if we find evidence of native pancreas insulin production, we will look at a variety of clinical variables to see if any correlate with recovery of function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included if:

Age greater than or equal to 18

GFR greater than 50 ml/min/1.73 m2

History consistent with T1DM prior to pancreas transplant

EXCLUSION CRITERIA:

Liver dysfunction (elevated liver enzymes, clinical evidence of portal hypertension)

coagulopathy (elevated INR or Partial Thromboplastin Time)

History of repeated instrumentation/cannulation in the jugular or femoral vessels

Dye allergy

Pregnancy

Known vascular anomalies

Anemia with Hgb less than 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-10-26; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Foulis AK, Liddle CN, Farquharson MA, Richmond JA, Weir RS. The histopathology of the pancreas in type 1 (insulin-dependent) diabetes mellitus: a 25-year review of deaths in patients under 20 years of age in the United Kingdom. Diabetologia. 1986 May;29(5):267-74. doi: 10.1007/BF00452061. PMID 3522324
- [Derived] Liu EH, Digon BJ 3rd, Hirshberg B, Chang R, Wood BJ, Neeman Z, Kam A, Wesley RA, Polly SM, Hofmann RM, Rother KI, Harlan DM. Pancreatic beta cell function persists in many patients with chronic type 1 diabetes, but is not dramatically improved by prolonged immunosuppression and euglycaemia from a beta cell allograft. Diabetologia. 2009 Jul;52(7):1369-80. doi: 10.1007/s00125-009-1342-7. Epub 2009 May 6. PMID 19418039